CLINICAL TRIAL: NCT00006115
Title: Alternation of FOLFOX6 (Oxaliplatin - Leucovorin - Fluorouracil) and FOLFIRI (Irinotecan - Leucovorin - Fluorouracil) as Second Line Treatment of Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068128; FRE-GERCOR-C98-3-FIREFOX; EU-20023
Record Dates: First submitted 2000-08-03; First posted 2004-03-08 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2002-01

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic colorectal cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of oxaliplatin, leucovorin calcium, and fluorouracil followed by irinotecan, leucovorin calcium, and fluorouracil in terms of progression free survival in patients with metastatic colorectal cancer. II. Evaluate these treatment regimens in terms of overall survival, response rate, toxicity, and quality of life in this patient population.

OUTLINE: This is a multicenter study. Patients receive 4 courses of oxaliplatin IV and leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours. Following the initial 4 courses of therapy, patients receive 4 courses of irinotecan IV over 30-90 minutes and leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Quality of life is assessed every 8 weeks. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 14-39 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the colon or rectum Measurable or evaluable lesion or residual disease (e.g., ascites, bone metastases) Failure after first line therapy Fluorouracil and leucovorin calcium OR Raltitrexed No oxaliplatin or irinotecan Relapse within 6 months of adjuvant therapy Relapse within 6 months of hepatic artery infusion chemotherapy for resected hepatic metastasis No symptomatic brain metastasis

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Hepatic: AST and ALT no greater than 3 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN Renal: Not specified Other: No bowel obstruction No other significant, uncontrolled underlying medical or psychiatric condition No serious active infection Neurologically stable No other prior malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix No psychological, social, familial, or geographical condition that would preclude study Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy Surgery: At least 2 weeks since prior surgery Other: No other concurrent experimental drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hebbar, MD, Study Chair — Centre Hospital Universitaire Hop Huriez
Locations (16):
- France (16):
  - Hopital Drevon, Dijon
  - Centre Jean Bernard, Le Mans
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - CH Meulan, Meulan-en-Yvelines
  - Intercommunal Hospital, Montfermeil
  - Centre Hospitalier de Mulhouse, Mulhouse
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Bichat-Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Hopital Claude Gallien, Quincy-sous-Sénart
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis
  - Clinique de l'Orangerie, Strasbourg